CLINICAL TRIAL: NCT05611814
Title: Preliminary Evaluation of an Osteopathic Manipulative Treatment (OMT) to Prevent Motion Sickness Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Aeromedical Research Laboratory (U.S. Federal Agency)
Collaborators: Alabama College of Osteopathic Medicine (Other); Department of Aviation Medicine, U.S. Army Medical Center of Excellence (Unknown)
Responsible Party: Principal Investigator, Amanda Kelley, Research Psychologist, United States Army Aeromedical Research Laboratory
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-019; M10996
Record Dates: First submitted 2022-11-01; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Between subjects design with two groups: sham and experimental (osteopathic manipulative treatment [OMT])
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants received treatment in private room. Study team and participants were blind to group (treatment received). Only the treatment administrator knew which treatment each participant received and was excluded from the remainder of the protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham treatment (Sham Comparator): The sham maneuver treatment addressed soft tissue tension, restriction of motion, and tenderness of the lower thoracic and lumbar regions.
  Interventions: Other: Sham treatment
- Experimental Osteopathic Manipulative Treatment (Experimental): The sham maneuver treatment addressed soft tissue tension, restriction of motion, and tenderness of the cervical region (targeted anatomical structures).
  Interventions: Other: Osteopathic Manipulative Treatment

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — Targeted anatomical structures are Scalene Muscles (Anterior/Middle/Posterior), Sternocleidomastoid Muscles (SCM), Suboccipital region, Cervical Paraspinal Muscles, Levator Scapulae Muscles, Upper Thoracic Paraspinal Muscles, Upper Trapezius Muscles, Atlanto-occipital (OA), Atlanto-axial (AA), C2-C7 vertebrae, T1-T4 vertebrae, Rib 1 bilaterally. Techniques include Suboccipital Myofascial Release, Soft tissue inhibition, kneading stretching, Facilitated Positional Release, and muscle energy technique.
  Arms: Experimental Osteopathic Manipulative Treatment
Other: Sham treatment — Targeted anatomical structures are Thoracic Paraspinal Muscles, Lumbar Paraspinal Muscles, Lower Trapezius Muscles, Sacrum, Supraspinatus, T5-T12, and Rib 2-12. Techniques include Soft tissue inhibition, Stretching, Kneading, counterstrain, Facilitated Positional Release, and muscle energy technique.
  L1-L5
  Arms: Sham treatment

SUMMARY:
Motion sickness directly impacts the readiness of the Army's aviation units. Severe motion sickness results in the dismissal of pilot and air crew candidates during initial training, while minor to moderate symptoms can be distracting during flight. The current medications on the market that target motion sickness symptoms are prohibited for use before flight. Osteopathic Manipulative Techniques are a low to no cost option, which lacks side effects, that allows Doctor of Osteopathic Medicine flight surgeons the opportunity to treat crew members without the use of pharmaceuticals. If effective, these techniques could be used to ensure aircrew readiness. Given the paucity of research on such a technique, a small, pilot study was conducted to demonstrate potential for such an approach.

ELIGIBILITY:
Inclusion Criteria:

* Must have normal hearing, vision or corrected to normal vision, and cognitive function as determined by self-report and review on demographics and personal history questionnaire.
* Must have obtained at minimum 6 hours of sleep prior to data collection, as assessed by self-report.
* Must have refrained from consumption of alcohol and Medications that impact motion sickness symptoms for a minimum of 16 hours prior to each test session, assessed by self-report.

Exclusion Criteria:

1. Must not be currently taking any medications that may affect the vestibular system as assessed by self-report and at the discretion of the study physician.
2. Must not have a history of vestibular disorders as assessed by self-report.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-24 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
Change in Motion sickness assessment questionnaire: gastrointestinal subscore from pre- to post-procedure | Administered immediately pre and post-procedure
  The Motion Sickness Assessment Questionnaire is a valid and reliable measure of the four dimensions of motion sickness: gastrointestinal, central, peripheral, and sopite-related (Gianaros, et al., 2001). It includes 16 items and response format is a likert scale (1 to 9). The difference in scores from pre- to post-procedure were calculated.
Change in Motion sickness assessment questionnaire: central subscore from pre- to post-procedure | Administered immediately pre and post-procedure
  The Motion Sickness Assessment Questionnaire is a valid and reliable measure of the four dimensions of motion sickness: gastrointestinal, central, peripheral, and sopite-related (Gianaros, et al., 2001). It includes 16 items and response format is a likert scale (1 to 9). The difference in scores from pre- to post-procedure were calculated.
Change in Motion sickness assessment questionnaire: peripheral subscore from pre- to post-procedure | Administered immediately pre and post-procedure
  The Motion Sickness Assessment Questionnaire is a valid and reliable measure of the four dimensions of motion sickness: gastrointestinal, central, peripheral, and sopite-related (Gianaros, et al., 2001). It includes 16 items and response format is a likert scale (1 to 9). The difference in scores from pre- to post-procedure were calculated.
Change in Motion sickness assessment questionnaire: sopite-related subscore from pre- to post-procedure | Administered immediately pre and post-procedure
  The Motion Sickness Assessment Questionnaire is a valid and reliable measure of the four dimensions of motion sickness: gastrointestinal, central, peripheral, and sopite-related (Gianaros, et al., 2001). It includes 16 items and response format is a likert scale (1 to 9). The difference in scores from pre- to post-procedure were calculated.
Change in Motion sickness assessment questionnaire: total subscore from pre- to post-procedure | Administered immediately pre and post-procedure
  The Motion Sickness Assessment Questionnaire is a valid and reliable measure of the four dimensions of motion sickness: gastrointestinal, central, peripheral, and sopite-related (Gianaros, et al., 2001). It includes 16 items and response format is a likert scale (1 to 9). The difference in scores from pre- to post-procedure were calculated.
Heart rate variability | Measured throughout procedure (10 minutes total)
  Heart rate was aggregated in 30-second intervals. Coefficients of variance were then calculated across the twenty 30-second intervals per participant.

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Aeromedical Research Laboratory, Fort Rucker, Alabama, United States

IPD SHARING:
Plan to Share IPD: No